CLINICAL TRIAL: NCT02905604
Title: Magnetic Stimulation of the Brain in Schizophrenia or Depression: A Randomized, Double Blind, Sham Controlled Trial of Repetitive Transcranial Magnetic Stimulation in Schizophrenia or Depression
Brief Title: Magnetic Stimulation of the Brain in Schizophrenia or Depression
Acronym: MA-SCH-DEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA-SCH-DEP
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia; Depression; Anhedonia; Avolition
Keywords: rTMS; negative symptoms; intermittent theta burst; iTBS; repetitive transcranial magnetic stimulation; dorsomedial prefrontal cortex; dmPFC; NIRS
MeSH Terms: conditions — Schizophrenia; Depression; Anhedonia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dmPFC iTBS (Experimental): Repetitive transcranial magnet stimulation (rTMS) over the dorsomedial prefrontal cortices at 90% of the resting motor threshold of the foot flexors. The rTMS is given in 20 trains to the left and right dmPFC, respectively. Each train consists of 10 bursts at 5 Hz (theta-frequency), and each burst consists of 3 pulses at 50 Hz. The stimulation is intermittent with 2 seconds of stimulation, 8 seconds off. After a 15 minute break the whole protocol i applied again, resulting in 2400 pulses/day. Treatment is delivered daily at 10 week days.
  Interventions: Device: dmPFC iTBS
- dmPFC Sham iTBS (Sham Comparator): A sham treatment protocol by using a sham coil with two identical sides where one side give active treatment as described above while on the other side the coil is insulated so very little magnetic energy is delivered. The coil has a built in positioning sensors and a software handling the randomization codes prompts the operator which side of the coil that should be directed towards the patient. Superficial transcutaneous electrical nerve stimulation (TENS) is applied over the stimulation site of the dmPFC synchronous wiht the TMS pulses to further mimic the sensation of the active stimulation.
  Interventions: Device: dmPFC Sham iTBS

INTERVENTIONS:
Device: dmPFC iTBS — 2400 pulses/day over 10 week days over bilateral dmPFC using MagPro X100 and the cool D-B80 A/P coil
  Other Names: rTMS with intermittent theta-burst frequency
  Arms: dmPFC iTBS
Device: dmPFC Sham iTBS — Sham iTBS
  Arms: dmPFC Sham iTBS

SUMMARY:
The primary objective is to evaluate if repetitive transcranial magnetic stimulation (rTMS) with theta burst frequency over dorsomedial prefrontal cortex (DMPFC) is an effective treatment for negative symptoms (anhedonia and avolition) in schizophrenia or depression. Other objectives are to increase the understanding of the underlying neurobiology of negative symptoms and the mechanisms for the treatment effect of rTMS.

DETAILED DESCRIPTION:
This is a double blind parallel randomized sham controlled trial. The intervention is intermittent theta-burst stimulation (iTBS), which is rTMS with theta burst frequency with 2400 pulses/day in two sessions at 90% of resting motor threshold intensity over the DMPFC, given in ten days on week days (10 treatment days must be completed within a maximum of 21 days). Stratified (depression and schizophrenia diagnosis) block randomization will be used for treatment allocation to active or sham side of the stimulation coil.

Patients will be referred from their regular psychiatric care facilities. At the screening visit the patient will be assessed if fulfilling all inclusion and none of the exclusion criteria. At the baseline visit thorough psychiatric, cognitive and neurophysiological examination will be performed. The latter include investigation of cortical excitability with paired-pulse TMS, mismatch negativity (MMN, a measure of aberrant stimulus detection), startle-response, habituation, electrodermal activity (EDA), near-infrared spectroscopy (NIRS), 24 hour actigraphy and heart rate registration.

During 10 week days the participants will receive a daily rTMS (or sham) treatment. On the day after last rTMS treatment the examinations performed at the baseline visit will be repeated. Four weeks after baseline there is a shorter visit to follow-up symptoms and functioning. At the end of this visit the blinding is unmasked and patients who have received sham rTMS will be offered active treatment in an open-phase. After the four weeks follow-up there are two additional and identical visits at 10 and 26 weeks after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia spectrum disorders or uni- or bipolar depression verified through a Mini International Neuropsychiatric Interview (M.I.N.I.)
* negative symptoms with anhedonia and avolition: ≤40 points on the The Motivation and Pleasure Scale-Self-Report (MAP-SR)
* unchanged medication the past month
* provision of signed informed consent form

Exclusion Criteria:

* epilepsy
* conductive ferromagnetic or other magnetic sensitive metals implanted in the head or within 30 cm of the treatment coil
* implanted device that is activated or controlled in any way by physiological signals
* implanted mediation pumps
* intracardiac lines, even when removed
* addiction (illicit drugs or alcohol) and pregnancy
* any condition that seriously increases the risk of non-compliance or loss of follow-up

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Mean change of total score on the Clinical Assessment Interview for Negative Symptoms (CAINS). | From baseline to day after last treatment, i.e. 14-21 days after baseline

SECONDARY OUTCOMES:
Mean change of total score on the CAINS | From baseline to four weeks after baseline.
Change in Clinical Global Impression (CGI) score | From baseline to four weeks after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bodén, Ph.D, MD, Principal Investigator — Uppsala University
Locations (1):
- Department of neuroscience, psychiatry, unit for Brain Stimulation and psychiatric clinical trials, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malm E, Struckmann W, Persson J, Boden R. Pain trajectories of dorsomedial prefrontal intermittent theta burst stimulation versus sham treatment in depression. BMC Neurol. 2020 Aug 20;20(1):311. doi: 10.1186/s12883-020-01881-3. PMID 32819321